CLINICAL TRIAL: NCT01572012
Title: Phase 1 Open-Label Randomized 4 Period Crossover Study Comparing Safety, Tolerability and PK of Ondansetron Given Subcutaneously With Hylenex Recombinant and Given Alone Intramuscularly, Intravenously and Orally in Healthy Volunteers
Brief Title: Phase 1 Safety, Tolerability and PK Study of Ondansetron and Hylenex Recombinant in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HALO-102-102
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety; Healthy Volunteers; tolerability
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subcutaneous Administration (Experimental): Ondansetron + Hylenex administered subcutaneously
  Interventions: Drug: Ondansetron + Hylenex
- Oral Administration (Experimental): Ondansetron administered orally
  Interventions: Drug: Zofran ODT
- Intramuscular Administration (Experimental): Ondansetron administered intramuscularly
  Interventions: Drug: Ondansetron
- Intravenous Administration (Experimental): Ondansetron administered intravenously
  Interventions: Drug: Ondansetron solution

INTERVENTIONS:
Drug: Ondansetron — Ondansetron solution 4 mg single administration
  Other Names: Zofran
  Arms: Intramuscular Administration
Drug: Ondansetron + Hylenex — Ondansetron solution (4 mg) single administration + Hylenex recombinant (150 U) single administration
  Other Names: Zofran
  Arms: Subcutaneous Administration
Drug: Zofran ODT — Zofran ODT (8 mg) single administration
  Other Names: ondansetron disintegrating tablet - oral
  Arms: Oral Administration
Drug: Ondansetron solution — Ondansetron solution (4 mg) single administration
  Other Names: Zofran
  Arms: Intravenous Administration

SUMMARY:
This is a randomized, open-label Phase 1 pharmacokinetic, tolerability, and safety study of ondansetron and Hylenex given subcutaneously compared to ondansetron given intravenously, intramuscularly, and orally in normal healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, open label, 4 way crossover Phase 1 study of the pharmacokinetics, safety and tolerability of a 4 mg dose of ondansetron administered subcutaneously with Hylenex recombinant compared to 4 mg doses of ondansetron administered intravenously and intramuscularly and an 8 mg dose of ondansetron administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 19-65 years old
* Females must be nonlactating and nonpregnant (negative serum pregnancy test at screening)and agree to practice effective birth control for at least 30 days after study completion
* Nonsmoker or no tobacco/nicotine use in previous 6 months
* Intact normal skin without obscuring tattoos, pigmentation or lesions
* Adequate venous access in upper extremities
* Normal vital signs, ECG, and labs or assessed by the Investigator as NCS
* Serum hemoglobin within site's normal range
* Negative drug and alcohol screen
* Able to make decisions and comply with study requirements

Exclusion Criteria:

* History of drug or alcohol abuse or positive drug and alcohol screen
* Abdominal surgery within the last 30 days
* Phenylketonuria
* Tobacco or nicotine use within previous 6 months
* Hypersensitivity or contraindication to ondansetron or other 5-HT3 receptor agonists
* Received ondansetron within 4 days prior to Day 1
* Known allergy to hyaluronidase or other ingredient in Hylenex recombinant
* Lower extremity edema
* Creatinine clearance < 60 mL/min
* Dehydration (Grade 2 or higher)
* Hypersensitivity or contraindication to heparin
* Abnormal ECG with clinically significant QT prolongation or history of
* Female who is pregnant or breastfeeding
* Participation in a clinical trial (drug or device) within 30 days of enrollment
* Clinically significant medical history, major systemic disease, intercurrent illness, physical examination finding, or clinical laboratory test result that risks the subject's safety or interfere with interpretation of study results
* Not able to comply with study requirements

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of Overall Safety | Days 1-31
  Investigator assessment of infusion site observations for parenteral administration; Subject assessment of pain using the verbal response scale for parenteral administration; Subject assessment of pain using the visual analog scale for parenteral administration; Investigator assessment of systemic adverse events

SECONDARY OUTCOMES:
Evaluation of Pharmacokinetics | Days 1-5
  Area of under the plasma concentration time curve (AUC); Time to achieve maximum plasma concentration (tmax); Maximum plasma concentration (Cmax); Plasma elimination half-life (t1/2); Relative bioavailability, ondansentron SC with Hylenex recombinant relative to ondansetron alone IV, IM, and PO

CONTACTS AND LOCATIONS:
Overall Officials: Samuel S Dychter, MD, Study Director — Halozyme Therapeutics
Locations (1):
- Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- [Derived] Dychter SS, Harrigan R, Bahn JD, Printz MA, Sugarman BJ, DeNoia E, Haughey DB, Fellows D, Maneval DC. Tolerability and pharmacokinetic properties of ondansetron administered subcutaneously with recombinant human hyaluronidase in minipigs and healthy volunteers. Clin Ther. 2014 Feb 1;36(2):211-24. doi: 10.1016/j.clinthera.2013.12.013. Epub 2014 Jan 31. PMID 24486335